CLINICAL TRIAL: NCT07380100
Title: Development of a Qualitative Scale to Asses the Acceptability of Percutaneous Techniques. A Delphi Study
Acronym: Accept_scale
Status: Active, not recruiting | Type: Observational
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Alberto Carcasona Otal, Principal Investigator, Universidad de Zaragoza
Other Study IDs: Acceptability Scale
Record Dates: First submitted 2026-01-13; First posted 2026-02-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Acceptability of Percutaneous Interventions
Keywords: Acceptability; Scale; Percutaneous Interventions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experts Panel: 20 experts (3 women and 17 men) took part in the study. The expert panel consisted of 14 physiotherapists, 2 psychologists, and 3 physicians
  Interventions: Other: Iterative focus group sessions and individual evaluation phases

INTERVENTIONS:
Other: Iterative focus group sessions and individual evaluation phases — The expert panel conducted iterative focus group sessions and successive individual evaluation phases until consensus was reached on the development of the acceptability scale.

SUMMARY:
This study aims to develop a new evaluation tool to assess patient acceptability of percutaneous interventions. A Delphi methodology will be implemented, involving the recruitment of a panel of experts in percutaneous interventions and pain management. The scale will be developed through several iterative phases until a final version is reached, comprising clearly defined domains, subdomains, items, and questions to be answered by patients in order to obtain an overall acceptability score for the percutaneous technique received. The scale is intended to be applicable across a wide range of percutaneous interventions and, consequently, to a broad patient population undergoing different percutaneous treatments depending on their clinical condition.

DETAILED DESCRIPTION:
This study aims to develop a new evaluation tool to assess patient acceptability of percutaneous interventions. A Delphi methodology will be implemented, involving the recruitment of a panel of experts in percutaneous interventions and pain management. The scale will be developed through several iterative phases until a final version is reached, comprising clearly defined domains, subdomains, items, and questions to be answered by patients in order to obtain an overall acceptability score for the percutaneous technique received. The scale is intended to be applicable across a wide range of percutaneous interventions and, consequently, to a broad patient population undergoing different percutaneous treatments depending on their clinical condition.

ELIGIBILITY:
Experts were required to:

* have at least five years of experience in percutaneous techniques
* have clinical experience working with patients with pain

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Experts in percutaneous interventions and pain management
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Consensus among the experts | Consensus will be achieved through 5 evaluation phases: Day 1 after first focus group Day 7 after second focus group Month 1 after first individual evaluation Month 2 after second individual evaluation Month 4 after second individual evaluation
  Consensus must be achieved among the experts panel to establish final decisions on the acceptability scale development.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zaragoza, Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on a reasonable request contacting with the main author once data has been published.
  Anyway, Individual participant data (IPD) will be shared with other researchers in accordance with data sharing protocols and participant consent, ensuring confidentiality and ethical considerations are maintained.
Supporting Information: Study Protocol, SAP
Time Frame: Once research has been published
Access Criteria: Study protocol will be publish in a scientific journal.